CLINICAL TRIAL: NCT01897480
Title: A Randomized, Controlled Phase 2 Study Evaluating LY2875358 Plus Erlotinib Versus Erlotinib as First-Line Treatment in Metastatic Non-Small Cell Lung Cancer Patients With Activating EGFR Mutations Who Have Disease Control After an 8-Week Lead-In Treatment With Erlotinib
Brief Title: A Study of LY2875358 in Participants With Non-Small Cell Lung Cancer With Activating Epidermal Growth Factor Receptor Mutations
Acronym: Balise
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14209; I4C-MC-JTBB (Other: Eli Lilly and Company); 2024-514268-18-00 (EU CTIS Number)
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — emibetuzumab; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2875358 plus Erlotinib (Experimental): Lead In: Approximately 8 weeks of erlotinib 150 milligram (mg) given orally per day.
  Randomization: Erlotinib 150 mg given orally per day plus 750 mg LY2875358 given as 1.5 hours intravenous (IV) infusions on Days 1 and 15 of 28-day cycles.
  Interventions: Biological: LY2875358; Drug: Erlotinib
- Erlotinib (Active Comparator): Lead In: Approximately 8 weeks of erlotinib 150 mg given orally per day.
  Randomization: Continue Erlotinib 150 mg given orally per day, in 28-day cycles.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Biological: LY2875358 — Administered IV
  Arms: LY2875358 plus Erlotinib
Drug: Erlotinib — Administered Orally

SUMMARY:
The primary purpose of this study is to compare the efficacy of the study drug LY2875358, given together with erlotinib, against erlotinib, alone. Participants will have Non-Small Cell Lung Cancer (NSCLC) that has advanced to Stage IV. Participants should not have been treated with drugs for Stage IV NSCLC, previously. All participants will get erlotinib alone, for approximately 8 weeks. Participants with radiographic disease control at the end of the erlotinib lead-in study period will be randomly assigned to receive LY2875358 plus erlotinib or erlotinib alone. Participants, who were chosen to receive erlotinib, alone, may cross over to the combination treatment at the time of progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of metastatic Stage IV NSCLC
* Have at least 1 measurable lesion whose presence is assessable using standard techniques by Response Evaluation Criteria in Solid Tumors (RECIST version 1.1)
* Have molecular evidence of an epidermal growth factor receptor mutation (EGFRmt) known to be associated with EGFR tyrosine kinase inhibitor (TKI) drug sensitivity (G719X, exon 19 deletion, L858R, L861Q)
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Haven't received any prior systemic chemotherapy for Stage IV NSCLC (unless received as neoadjuvant or adjuvant therapy for early-stage NSCLC disease and completed therapy at least 6 months prior to enrollment)
* Availability of adequate tumor material (block or slides)

Exclusion Criteria:

* Are currently enrolled in, or discontinued within the last 30 days from, a clinical trial involving an investigational product or non-approved use of a drug or device
* Have previously completed or withdrawn from this study or any other study investigating LY2875358
* Have a serious concomitant systemic disorder or significant cardiac disease
* Have interstitial pneumonia or interstitial fibrosis of the lung or have pleural effusion, pericardial fluids or ascites, requiring drainage every other week or more frequently
* Have a history of another malignancy except for basal or squamous cell skin cancer and/or in situ carcinoma of the cervix, or other solid tumors treated curatively and without evidence of recurrence for at least 3 years prior to the study
* Have major surgery less than 2 weeks prior to the initiation of study treatment therapy
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2013-08-28 (Actual); Primary Completion 2016-03-14 (Actual); Study Completion 2026-01-08 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Randomization to Objective Disease Progression or Death Due to Any Cause (Estimated 3 Years)

SECONDARY OUTCOMES:
Change in Tumor Size (CTS) | Baseline to Measurement with Smallest Tumor Size (Estimated 3 Years)
Proportion of Participants Exhibiting a Confirmed Complete Response (CR) or Partial Response (PR) (Overall Response Rate [ORR]) | Baseline to Objective Disease Progression or Start of New Anticancer Therapy (Estimated 3 Years)
Duration of Response (DoR) | Date of CR or PR to Date of Objective Disease Progression or Death Due to Any Cause (Estimated 3 Years)
Time to Progressive Disease (TTPD) | Randomization to Objective Disease Progression (Estimated 3 Years)
Proportion of Participants Exhibiting a Stable Disease (SD) or a confirmed CR or PR (Disease Control Rate [DCR]) | Baseline to Objective Disease Progression or Participant Stops Study (Estimated 3 Years)
Overall Survival (OS) | Randomization to Death Due to Any Cause (Estimated 5 Years)
Change from Baseline in European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaires (QLQ) C30 (QLQ-C30) and Lung Cancer 13 (QLQ-LC13) | Baseline, Objective Disease Progression or Participants Stops Study (Estimated 3 Years)
Pharmacokinetics (PK): Area Under the Concentration Time Curve During a Dosing Interval (AUCtau) of LY2875358 and Erlotinib | Baseline through Cycle 4 (28 Day Cycle)
Proportion of Participants with Anti-LY2875358 Antibody Response | Baseline through 30 Day Follow Up (Estimated 3 Years)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (45):
- Denmark (3):
  - Herlev and Gentofte Hospital, Herlev, Capital Region
  - Rigshospitalet, Copenhagen, Copenhagen
  - Odense Universitetshospital, Odense C, Syd
- France (6):
  - CHU de Caen Hopital Cote de Nacre, Caen
  - Chu Gabriel Montpied, Clermont-Ferrand
  - CHU De Grenoble Hopital Albert Michallon, Grenoble
  - HCL-Hôpital Louis Pradel, Lyon (Bron) Cedex
  - Hôpital Arnaud de Villeneuve - CHU Montpellier, Montpellier
  - CHU la Miletrie, Poitiers
- Germany (6):
  - Klinik Schillerhöhe, Gerlingen, Baden-Wurttemberg
  - Thoraxklinik-Heidelberg gGmbH, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Klinikum Köln-Merheim, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Helios Klinikum Emil von Behring Berlin-Zehlendorf, Berlin
- Italy (5):
  - Azienda Ospedaliera Universitaria Careggi, Florence, Florence
  - Azienda Sanitaria Ospedaliera S Luigi Gonzaga, Orbassano, Torino
  - Istituto Oncologico Veneto IRCCS, Padua, Veneto
  - Istituto Tumori ""Giovanni Paolo II, Bari
  - Istituti Ospedalieri di Cremona, Cremona
- Netherlands (4):
  - Jeroen Bosch Hospital, 's-Hertogenbosch, North Brabant
  - Ziekenhuis Rijnstate, Arnhem
  - Ziekenhuis St. Jansdal, Harderwijk
  - St. Antonius Ziekenhuis, locatie Nieuwegein, Nieuwegein
- South Korea (7):
  - Chungbuk National University Hospital, Cheongju-si, Chungcheongbuk-do [Chungbuk]
  - Gachon University Gil Medical Center, Namdong-gu, Incheon-gwangyeoksi [Incheon]
  - Severance Hospital, Yonsei University Health System, Seoul, Korea
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Ulsan University Hospital, Ulsan, Ulsan-Kwangyǒkshi
- Spain (5):
  - Corporacion Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Puerta De Hierro, Majadahonda, Madrid
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Clinica Universitaria De Navarra, Pamplona, Navarre
  - Hospital del Mar, Barcelona
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (5):
  - Gartnavel General Hospital, Glasgow, Glasgow City
  - Charing Cross Hospital, Chelsea, London
  - Wythenshawe Hospital, Wythenshawe, Manchester
  - New Cross Hospital, Wolverhampton, West Midlands
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/